CLINICAL TRIAL: NCT07274930
Title: Effect of Gluten-free Casein-free Diet on Serum Zonulin and Claudin-5 Levels and Some Clinical Symptoms in Children With Autism Spectrum Disorder: A Randomized Controlled Trial
Brief Title: Effect of Gluten-free Casein-free Diet on Serum Zonulin and Claudin-5 Levels and Some Clinical Symptoms in Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Elif Ozturk, Research Assistant (PhD Student), Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 223S497
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Autism Spectrum Disorder (ASD); Nutrition
Keywords: autism specktrum disorder; gluten-free casein-free diet; intestinal permeability; zonulin; claudin-5
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gluten Free Casein Free Diet (Experimental): The group following a ASD
  Interventions: Other: Gluten Free Casein Free Diet
- Normal Diet (Active Comparator): Normal Diet
  Interventions: Other: Normal Diet

INTERVENTIONS:
Other: Gluten Free Casein Free Diet — Gluten Free Casein Free Diet
  Arms: Gluten Free Casein Free Diet
Other: Normal Diet — Participants follow a normal diet
  Arms: Normal Diet

SUMMARY:
This study will investigate the effects of a gluten-free casein-free diet (GFCF) on serum zonulin and claudin-5 levels in children diagnosed with ASD, in relation to intestinal permeability and blood-brain barrier permeability, and on electroencephalography (EEG) findings, autism symptoms, and some clinical symptoms. The study also included EEG findings to measure brain cortical activity in children diagnosed with autism before and after the diet.

Purpose:

This study aimed to investigate the effects of the GFCF dietary model on serum zonulin and claudin-5 levels, autism spectrum disorder parameters, gastrointestinal symptoms, and some clinical symptoms.

Objectives:

1. Examination of serum zonulin and claudin-5 levels in the GFCF group compared to the control group.
2. Examination of EEG findings in the GFCF group compared to the control group.
3. Examination of Childhood Autism Assessment Scale scores in the GFCF group compared to the control group.
4. Examination of Autism Behavior Checklist scores in the GFCF group compared to the control group.
5. Examination of gastrointestinal sensitivity index scores in the GFCF group compared to the control group.
6. Examination of the diet quality index in individuals diagnosed with GFCF at the end of the study.

Participants:

This study will be conducted on children aged 3-6 years who were initially diagnosed and who had not used any nutritional supplements and/or medications and who had not followed any diet.

Inclusion criteria:

Children diagnosed with ASD will undergo general examinations by a pediatric neurologist, psychiatrist, and dietitian, and eligible participants will be included in the study. All children will be evaluated by a child and adolescent psychiatrist according to DSM-5 diagnostic criteria, and all will have their neurological evaluations completed by a pediatric neurologist. Children diagnosed with autism spectrum disorder who receive at least two hours of regular special education per week will be included in the study.

Special education is crucial for every child diagnosed with ASD. The project team considers the importance of special education for children with ASD. It has been stated that participants who do not receive special education or are not continuing their education will be excluded. However, children's special education hours vary widely. The state provides two hours of special education for diagnosed children. Further hours of education may vary based on family requests. Because each child in this study will be evaluated after three months based on their individual development, it is expected that their education hours will remain constant throughout the study. If each participating child receives two hours of special education during the study, the continuity of these two hours will be monitored. If a change in training hours is detected, participants will be excluded from the study. Analysis will be conducted by adjusting for the effect of training hours to determine the effect of the diet.

Individuals who meet the study criteria and voluntarily agree to participate in the study will be provided with an informed consent form. The Childhood Autism Rating Scale (CARS) and the Problem Behavior Checklist (ABC) will be used in the clinical evaluation of all children. These scales will be completed by the same clinician during the initial psychiatric evaluation and immediately after completing the 12-week diet program.

Blinding will be applied to the CARS, ABC, gastrointestinal sensitivity index, Bristol stool scale, and serum zonulin and claudin-5 analyses administered to the participants at the beginning and end of the study. Except for the dietitian researcher responsible for explaining and monitoring the nutrition education and diet plan, all other researchers will evaluate the participants in accordance with the blinding principle.

Exclusion criteria:

Those under three years of age and over six years of age; Those unable to be fed orally; Patients with height-for-age, weight-for-age, and BMI-for-age Z scores above +2 SD and below -2 SD for their age and gender using World Health Organization growth references; those diagnosed with neurometabolic diseases such as epilepsy, Fragile X syndrome, or Williams syndrome; those who do not continue their special education or do not accept special education; those who are on any dietary treatment, using nutritional supplements and/or medication in the last 2 months; those with diet compliance less than 80%; and those diagnosed with celiac disease and gluten intolerance will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

Children diagnosed with ASD will undergo general examinations by a pediatric neurologist, psychiatrist, and dietitian, and eligible participants will be included in the study. All children will be evaluated by a child and adolescent psychiatrist according to DSM-5 diagnostic criteria, and all will have their neurological evaluations completed by a pediatric neurologist. Children diagnosed with autism spectrum disorder who receive at least two hours of regular special education per week will be included in the study.

Special education is crucial for every child diagnosed with ASD. The project team considers the importance of special education for children with ASD. It has been stated that participants who do not receive special education or are not continuing their education will be excluded. However, children's special education hours vary widely. The state provides two hours of special education for diagnosed children. Further hours of education may vary based on family requests. Because each child in this study will be evaluated after three months based on their individual development, it is expected that their education hours will remain constant throughout the study. If each participating child receives two hours of special education during the study, the continuity of these two hours will be monitored. If a change in training hours is detected, participants will be excluded from the study. Analysis will be conducted by adjusting for the effect of training hours to determine the effect of the diet.

Individuals who meet the study criteria and voluntarily agree to participate in the study will be provided with an informed consent form. The Childhood Autism Rating Scale (CARS) and the Problem Behavior Checklist (ABC) will be used in the clinical evaluation of all children. These scales will be completed by the same clinician during the initial psychiatric evaluation and immediately after completing the 12-week diet program.

Blinding will be applied to the CARS, ABC, gastrointestinal sensitivity index, Bristol stool scale, and serum zonulin and claudin-5 analyses administered to the participants at the beginning and end of the study. Except for the dietitian researcher responsible for explaining and monitoring the nutrition education and diet plan, all other researchers will evaluate the participants in accordance with the blinding principle.

Exclusion Criteria:

Those under three years of age and over six years of age; Those unable to be fed orally; Patients with height-for-age, weight-for-age, and BMI-for-age Z scores above +2 SD and below -2 SD for their age and gender using World Health Organization growth references; those diagnosed with neurometabolic diseases such as epilepsy, Fragile X syndrome, or Williams syndrome; those who do not continue their special education or do not accept special education; those who are on any dietary treatment, using nutritional supplements and/or medication in the last 2 months; those with diet compliance less than 80%; and those diagnosed with celiac disease and gluten intolerance will be excluded from the study.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
The effect of the GFCF diet on blood zonulin level | 3 months
  The effect of the GFCF diet on blood zonulin level
The effect of the GFCF diet on blood claudin-5 level | 3 months
  The effect of the GFCF diet on blood claudin-5 level

CONTACTS AND LOCATIONS:
Overall Officials: Aslı Akyol, Study Chair — Hacettepe Univercity
Locations (1):
- Karadeniz Teknik Üniversitesi, Trabzon, Ortahi̇sar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: The Efficacy of the Gluten-free Case in-free Diet for Moroccan Autistic Children — https://www.foodandnutritionjournal.org/volume6number3/the-efficacy-of-the-gluten-free-case-in-free-diet-for-moroccan-autistic-children/
- See also: Serum zonulin level in autistic children and its relation to severity of symptoms a case-control study — https://www.nature.com/articles/s41598-025-11420-0